CLINICAL TRIAL: NCT01232894
Title: A 12 Week, Multi-center, Randomized, Open Label Study, eValuating the Efficacy and Safety of Treatment Regimens That Include ONbrez (Indacaterol) in Patients With Moderate to Severe COPD (MOVE-ON Study)
Brief Title: 12-week Open-label Evaluation of Efficacy and Safety of Indacaterol
Acronym: MOVE-ON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149BIL01
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: indacaterol; COPD; Long-acting beta2-agonist (LABA)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol (Experimental): Indacaterol 150 µg once-daily via single-dose dry powder inhaler
  Interventions: Drug: Indacaterol
- Long-acting beta2-agonist (Active Comparator): Participants' current long-acting beta2-agonist (LABA) bronchodilator therapy
  Interventions: Drug: Long-acting beta2-agonist

INTERVENTIONS:
Drug: Indacaterol — Indacaterol 150 µg once-daily via single-dose dry powder inhaler
  Arms: Indacaterol
Drug: Long-acting beta2-agonist — Long-acting beta2-agonist (LABA) bronchodilator monotherapy via inhaler twice daily
  Arms: Long-acting beta2-agonist

SUMMARY:
In this 12-week study, patients were randomized to either open-label indacaterol or standard of care for Chronic Obstructive Pulmonary Disease (COPD) treatment; efficacy and safety were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2007) and:
* Post-bronchodilator forced expiratory volume in 1 second (FEV1) <80% and ≥30% of the predicted normal value
* Post-bronchodilator FEV1/FVC (Forced Vital Capacity) <70%
* Current COPD bronchodilator treatment that includes a LABA bronchodilator or a fixed dose combination of LABA and Inhaled Corticosteroid (ICS)

Exclusion Criteria:

* Patients with a history of asthma
* Patients who are currently being treated for COPD with tiotropium (Spiriva®)
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Israel (8):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Holon
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 90 participants were screened and enrolled into the study. The participants were randomized in a 2:1 ratio. Out of 90 participants randomized, 87 received study drug and were included in the Safety set for analysis.
Period: Overall Study
Arm/Group | Indacaterol | Long-acting beta2-agonist
Started | 60 | 30
Received Study Drug | 59 | 28
Completed | 48 | 22
Not Completed | 12 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 8 | 5
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol | Long-acting beta2-agonist | Total
Number analyzed (Participants) | 60 | 30 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.9) | 64.8 (9.9) | 65.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 46 | 20 | 66

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on Clinical COPD Questionnaire (CCQ) Score
Description: The Clinical Chronic Obstructive Pulmonary disease (COPD) Questionnaire (CCQ) is a self-administered questionnaire containing ten questions, divided into three domains: symptoms, mental and functional state. The questions are based on a 7-point scale where a '0' means having no limitations and a '6' means extreme or complete limitations. The final score is the mean of all ten questions. The CCQ score was recalculated according to the paper by Van der Molen et al., 2003. The statistical significance remained the same.
Time Frame: Baseline and 12 weeks
Population: Full analysis Set: all patients who received at least one dose of study drug and have evaluable data for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Indacaterol | Long-acting beta2-agonist
Number analyzed (Participants) | 55 | 24
units on a scale
  Baseline | 1.8 (1.0) | 1.7 (0.7)
  12 weeks | 1.7 (1.1) | 1.9 (1.0)

ADVERSE EVENTS:
Time Frame: Entire duration of study
Description: Out of 90 participants randomized, 87 received study drug and were included in the safety set for analysis.
Arm/Group | Indacaterol | Long-acting beta2-agonist
Serious Adverse Events (participants affected / at risk) | 3/59 | 0/28
Other Adverse Events (participants affected / at risk) | 9/59 | 4/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indacaterol (N=59) | Long-acting beta2-agonist (N=28)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indacaterol (N=59) | Long-acting beta2-agonist (N=28)
Dizziness (Nervous system disorders) | 3 (4) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.